CLINICAL TRIAL: NCT07143695
Title: Parasternal Intercostal Muscle Thickening as an Additive Weaning Criterion to Minimize Re-intubation Rate: a Randomized Controlled Trial
Brief Title: Parasternal Intercostal Muscle Thickening as an Additive Weaning Criterion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mina Adolf Helmy, Lecturer of anesthesia and critical care, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PIC criterion
Record Dates: First submitted 2025-08-20; First posted 2025-08-27 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Critically Ill
Keywords: Weaning; re-intubation; mechanical ventilation
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Sham Comparator): patients in control will be weaning using standard criteria
  Interventions: Device: Sham parasternal intercostal thickening
- Ultrasound (Active Comparator): patient in this group will be weaned using standard criteria plus mean parasternal thickening fraction less than 6.5 %
  Interventions: Device: Parasternal intercostal thickening fraction

INTERVENTIONS:
Device: Parasternal intercostal thickening fraction — Parasternal intercostal thickening fraction less than 6.5%
  Arms: Ultrasound
Device: Sham parasternal intercostal thickening — Ultrasound assessment only for purpose of blinding
  Arms: Control group

SUMMARY:
Increased days of MV are not without hazards, including barotraumas and ventilator-associated pneumonia. Similarly, premature separation of MV is associated with increased mortality secondary to adverse cardiorespiratory events. Therefore, the time of weaning should be wisely evaluated. There is growing evidence concerning respiratory muscles dysfunction that contributes to difficulty or prolonged liberation from MV.

DETAILED DESCRIPTION:
Researchers aim to evaluate the influence of adding parasternal thickening fraction to the standard weaning criteria and its impact on reintubation

ELIGIBILITY:
Inclusion Criteria:

* critically ill patient mechanically ventilated for 24 hours or more first spontaneous breathing trial

Exclusion Criteria:

* patient refusal difficult ultrasound views tracheostomized patient neuromuscular disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of reintubation | Within 72 hours after extubation
  need for reintubation

SECONDARY OUTCOMES:
Incidence of weaning failure | within 72 hours post-extubation
  failed spontaneous breathing trial or reintubation

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
IPD might not be shared to protect confidentiality, maintain competitive advantage, and comply with legal or contractual restrictions

REFERENCES:
- [Background] Helmy MA, Hasanin A, Milad LM, Mostafa M, Fathy S. Parasternal intercostal muscle thickening as a predictor of non-invasive ventilation failure in patients with COVID-19. Anaesth Crit Care Pain Med. 2022 Jun;41(3):101063. doi: 10.1016/j.accpm.2022.101063. Epub 2022 Apr 26. No abstract available. PMID 35487407
- [Background] Helmy MA, Milad LM, Hasanin AM, Mostafa M, Mannaa AH, Youssef MM, Abdelaziz M, Alkonaiesy R, Elshal MM, Hosny O. Parasternal intercostal thickening at hospital admission: a promising indicator for mechanical ventilation risk in subjects with severe COVID-19. J Clin Monit Comput. 2023 Oct;37(5):1287-1293. doi: 10.1007/s10877-023-00989-4. Epub 2023 Mar 24. PMID 36961635
- [Background] Helmy MA, Hasanin A, Milad LM, Mostafa M, Hamimy WI, Muhareb RS, Raafat H. Ability of parasternal intercostal muscle thickening fraction to predict reintubation in surgical patients with sepsis. BMC Anesthesiol. 2024 Aug 22;24(1):294. doi: 10.1186/s12871-024-02666-8. PMID 39174907